CLINICAL TRIAL: NCT02337088
Title: Delayed Cord Clamping at 30 vs. 60 Seconds for Very Low Birth Weight Infants: A Randomized Controlled Trial
Brief Title: Delayed Cord Clamping in Very Low Birth Weight Infants
Acronym: DCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical reasons
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-0546
Record Dates: First submitted 2014-12-15; First posted 2015-01-13 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Very Low Birth Weight Infants; Premature Infants; Intraventricular Hemorrhage
Keywords: delayed cord clamping
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30 seconds (Active Comparator): For subjects in the 30 second arm, the umbilical cord will be clamped at 30 seconds after delivery.
  Interventions: Procedure: Delayed cord clamping at 30 seconds
- 60 seconds (Experimental): For subjects in the 60 second arm, the umbilical cord will be clamped at 60 seconds after delivery.
  Interventions: Procedure: Delayed cord clamping at 60 seconds

INTERVENTIONS:
Procedure: Delayed cord clamping at 30 seconds — For subjects enrolled in the 30 second arm, the umbilical cord will be clamped at exactly 30 seconds after delivery
  Arms: 30 seconds
Procedure: Delayed cord clamping at 60 seconds — For subjects enrolled in the 60 second arm, the umbilical cord will be clamped at exactly 60 seconds after delivery
  Arms: 60 seconds

SUMMARY:
The purpose of this study is to determine if there is a difference in neonatal outcomes with delayed umbilical cord clamping at 30 versus 60 seconds. Our primary outcome will be intraventricular hemorrhage (IVH) (bleeding in the brain) in these infants.

DETAILED DESCRIPTION:
Immediately following delivery, up to 40% of the total blood volume available to the infant is in the placenta. Over a period of 30 seconds to 3 minutes, a significant portion of this blood is transferred to the infant through the umbilical cord. Delayed cord clamping following delivery facilitates this transfer of blood.

Preterm infants are very susceptible to the effects of anemia and hypovolemia. A recent meta-analysis showed that a brief delay in umbilical cord clamping (30-60 seconds) decreases the risk of anemia, blood transfusion, intraventricular hemorrhage, necrotizing enterocolitis, and the need for blood pressure support after delivery. The same meta-analysis showed no impact on Apgar scores or hypothermia due to a brief delay in resuscitation efforts to allow delayed cord clamping.

Preterm infants are at significant risk for IVH and as high as 20% of very low birth weight infants will have it. IVH is an important cause of brain injury in these infants. In our study, we would like to determine the optimal timing of delayed cord clamping in order to prevent IVH in these infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are expected to deliver a very low birth weight infant
* Neonates born weighing >= 500g and <1500 grams
* Mother 18 years of age or older
* English speaking mother

Exclusion Criteria:

* Placental abruption
* Vasa previa
* Fetal hydrops or other signs of fetal volume overload
* Other major fetal anomalies
* Placenta Accreta
* Mother < 18 years of age
* Non-English speaking mother
* Infants >= 1500g (3.3 lbs) or <500g

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Intraventricular hemorrhage | During NICU admission up to 6 months
  Neonates will be followed for up to 6-months during NICU admission to assess for the development of intraventricular hemorrhage.

SECONDARY OUTCOMES:
Hemoglobin and hematocrit | During NICU admission up to 6 months
  Neonates will be followed for up to 6-months and initial H/H will be recorded.
Need for blood transfusion | During NICU admission up to 6 months
  Neonates will be followed for up to 6-months and assessed for clinical or laboratory evidence of need for transfusion.
Bilirubin levels | During NICU admission up to 6 months
  Neonates will be followed for up to 6-months and assessed for clinical jaundice.
Delivery room temperature | Delivery
  Neonates will be assessed for hypothermia at the time of delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States